CLINICAL TRIAL: NCT01772121
Title: Prevalence of Host and Viral Genotypes in Patients With Chronic Hepatitis B and Hepatitis C Infection in India
Brief Title: Observational Study on Prevalence of Host and Viral Genotypes in Chronic Hepatitis B and Hepatitis C Patients in India
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GX-US-174-0196
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis B; Hepatitis C
Keywords: HBV, HCV, chronic, India, observational study, prevalence,; genotypes, SNPs, viral hepatitis
MeSH Terms: conditions — Hepatitis B; Hepatitis C; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A portion of the blood drawn at the study visits will be frozen and stored. Stored blood samples may be used by the Sponsor or its research partners for HCV/HBV genotyping/phenotyping assays (as applicable) or their development or for retesting the amount of HCV/HBV in the blood. At the conclusion of this study, these samples may be retained in storage by Gilead Sciences or a designee for a period up to 10 years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HCV Cohort: A total of 1000 subjects were enrolled in the study and of that 500 subjects had a diagnosis of chronic HCV infection
- HBV Cohort: A total of 1000 subjects were enrolled in the study and of that 500 subjects had a diagnosis of chronic HBV infection

SUMMARY:
This study will define the substantial disease burden associated with viral hepatitis in India, and provide a foundation to understand the host and viral determinants of disease pathogenesis that may ultimately impact treatment decisions and outcome

DETAILED DESCRIPTION:
The overall goal of this study is to correlate the host and viral genetics of patients infected with viral hepatitis with their clinical presentation. This study will provide the first nation-wide estimate of key host genetic polymorphisms associated with immune response, such as in the IL28B gene locus which has been associated with treatment outcomes in hepatitis C. Characterization of HCV and HBV viral genotypes and sub-types across different geographic regions will allow for an exploration of associations between host and viral genotypes. Another objective of this study is to identify co-morbid illness and metabolic factors that are associated with chronic liver disease due to viral hepatitis. Finally, this survey will explore patient awareness of their disease, risk factors for disease progression, and their treatment options

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Male or female, age >= 18
* Willing and able to comply with the visit procedure
* Prior diagnosis of chronic HCV infection or chronic HBV infection

Exclusion Criteria:

* History of difficulty with blood collection and/or poor venous access for the purposes of phlebotomy
* History of bleeding disorder
* Blood loss requiring transfusion or > 3 g/dL decrease in hemoglobin within 4 days of the visit
* Knowingly co-infected with HCV/HBV or with HIV
* Currently undergoing therapy for chronic hepatitis C or chronic hepatitis B
* Currently receiving treatment with any other investigational agent or device -- Enrolled in another clinical study evaluating a treatment or procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 1000 subjects will be enrolled in the study. Of these, it is planned that approximately 500 subjects will have a diagnosis of chronic HCV infection and approximately 500 subjects will have a diagnosis of chronic HBV infection.Subjects knowingly co-infected with HCV/HBV or HIV may not participate in the study
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Variation in the IL28B rs12979860 SNP | One Visit
  Characterize the variation in the IL28B rs12979860 SNP that exists among patients with chronic hepatitis C or chronic hepatitis B infection, in the different geographic regions of India

SECONDARY OUTCOMES:
Prevelance of HBV and HCV genotypes | One Visit
  Assess the prevalence of HBV and HCV genotypes and subtypes in different geographic regions of India
Characterize the SNPs present in innate immune factors toll-like receptor 7 (TLR7) | One Visit
  Characterize the SNPs present in innate immune factors TLR7 (rs3853839, rs179008); TLR9 (rs41308230, rs5743844 ); RIG-I (rs11795404, rs10813831) and NOD2 (rs2067085, rs2066842), in patients with chronic hepatitis C or chronic hepatitis B in the different geographic regions of India

CONTACTS AND LOCATIONS:
Locations (19):
- India (19):
  - Global Hospitals, Lakdi ka Pul, Hyderabad, Andhra Pradesh
  - Asian Institute of Gastroenterology , 6-3-661, Somajiguda, Hyderabad, Andhra Pradesh
  - Institute of digestive and liver disease,Ganeshguri, Guwahati, Assam
  - Liver Clinic, 203-204, Narmada Complex, Near Kadiwala School, Ring Road, Surat, Gujarat
  - Medanta-The Medicity,Sector - 38, Gurgaon, Haryana
  - Manipal Hospitals,98, HAL Airport Road, Bangalore, Karnataka
  - Diwaliben Mohanlal Mehta Charitable Trust ,1st Foor, Khatau Mansion,95/K Bhulabhai Desai Road, Mumbai, Maharashtra
  - Seth GS Medical College and KEM Hospital, Acharya Donde Marg, Parel, Mumbai, Maharashtra
  - Midas Institute of Gastro-enterology, Midas Height,7 - Central Bazar Road,Ramdaspeth, Nagpur, Maharashtra
  - Dharamsi Hospital,Chandni Chowk, South Shivajinagar, Sangli, Mahashtra
  - Civil Hospital, Dawrpui, Aizawl, Mizoram
  - Institute of Liver and Biliary Sciences, D-1, Vasant Kunj, New Delhi, New Delhi
  - Digestive Diseases Centre, Beam Diagnostics Premises, Bajrakabati Road [Mali Sahi], Bata Lane, Cuttack, Odhisa
  - Dayanand Medical College & Hospital, Tagore Nagar, Civil Lines, Ludhiana, Punjab
  - Rai Speciality Care Centre, H-6 Janpath,Shyamnagar,Ajmer Road, Sodala, Jaipur, Rajasthan
  - Global Hospitals & Health City,# 439, Cheran Nagar, Perumbakkam, Off OMR, Near Shollinganalur, Chennai, Tamil Nadu
  - VGM Hospital, 2100, Trichy Road, Rajalakshmi Mills Stop, Coimbatore, Tamil Nadu
  - Institute of Post Graduate Medical Education And Research,244 A.J.C Bose Road, Kolkata, West Bengal
  - Apollo Hospital, Seepat Road, Bilāspur